CLINICAL TRIAL: NCT00028145
Title: Perinatal Core Protocol
Brief Title: Prenatal and Postnatal Studies of Interventions for Prevention of Mother-To-Child Transmission
Status: Completed | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PACTG P1025; U01AI068632 (NIH)
Record Dates: First submitted 2001-12-13; First posted 2001-12-14 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: HIV Infections; Pregnancy Complications, Infectious
Keywords: Women's Health; Disease Transmission, Vertical; Preventive Medicine; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and amniotic fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Pregnant, HIV-infected women
  Interventions: Behavioral: Adherence assessment

INTERVENTIONS:
Behavioral: Adherence assessment — Adherence will be assessed using questionnaires at all study visits.

SUMMARY:
The purpose of this study is to collect and study clinical and laboratory information about a pregnant or new mother and her medical care that will increase our knowledge of the best care for HIV-infected pregnant women and their children.

The rate of transmission of HIV from mothers to their infants has gone down. Specific U.S. Public Health Service guidelines recommend that HIV-infected pregnant women be treated with anti-HIV therapies; but the effectiveness of treatment and safety for the mother and her infant have not been fully examined. This study will monitor the health of women and their infants while they receive anti-HIV therapy. Also, this study will provide information that may be used for future studies.

DETAILED DESCRIPTION:
The current low rate of vertical transmission of HIV in the U.S. limits the number and types of questions concerning transmission risk and pathogenesis that can be addressed by a single clinical trial. Specific U.S. Public Health Service guidelines recommend antiretroviral therapy (ART) during pregnancy to maximize health of women. However, data regarding the effectiveness and safety of and adherence to ART during pregnancy are limited. It is both appropriate and necessary for theInternational Maternal Pediatric Adolescent AIDS Clinical Trials Group (IMPAACT) to recruit pregnant women into a non-interventional, analytic, epidemiologic study to methodically collect clinical and laboratory data from them and their infants. This way, the IMPAACT can achieve the aims of evaluating management of HIV-infected women during pregnancy and determining the safety and effectiveness of ART and other interventions intended to prevent vertical transmission and/or improve maternal health. In addition, longitudinally collected core protocol data and repository specimens will enable future substudies.

Participants receive no protocol specific treatment or other intervention as part of this study. The study involves the follow-up of HIV-infected women enrolled during pregnancy or at the time of delivery for 6 months postpartum and their infants for the first 6 months of life. There will be 8 study visits for enrolled participants and 6 study visits for infants. Data concerning ART use, adherence to medications, and review of symptoms relevant to side effects and toxicities are collected through administration of questionnaires at all maternal visits. Phlebotomy is conducted to obtain specimens for a repository and for required laboratory tests. During labor and delivery, maternal blood is obtained for lymphocyte subset and viral load assays and for repository storage. Collection of amniotic fluid at the time of cesarean section is encouraged. These collections are submitted to a central repository. Data for the core protocol are abstracted from the infant's medical record at the time of birth and at each postnatal visit.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* At least 14 weeks pregnant OR have delivered a liveborn or stillborn infant and are within 14 days of the delivery
* Currently receiving care at an IMPAACT or other participating site
* Have a parent or guardian willing to provide signed informed consent, if applicable
* Mentally capable of giving informed consent to have the infant and self followed at an IMPAACT site

Exclusion Criteria:

* Intend to end the pregnancy
* Unable to come for a study visit within 14 days after delivery (if known to be HIV infected prior to delivery) OR within 28 days after delivery (if found to be HIV infected at the time of labor and delivery or within 14 days after delivery)

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinics
Sampling Method: Probability Sample
Enrollment: 3090 (Actual)
Dates: Start 2002-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Maternal and infant response to prescribed interventions | Throughout study
Immune and viral parameters of participants taking prescribed interventions | Throughout study

SECONDARY OUTCOMES:
Occurrences of genotypic and phenotypic resistance in HIV-infected mothers | Throughout study
Clinical, immunological, and virological responses in HIV-infected women | Throughout study
Mother-to-child transmission rates of resistance mutations | Throughout study
Adherence to ART among HIV-infected pregnant women during pregnancy and postpartum | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Tuomala, MD, Study Chair — Director of Obstetrics and Gynecology, Brigham and Women's Hospital; Gwen Scott, MD, Study Chair — Pediatric Infectious Diseases, University of Miami School of Medicine
Locations (77):
- United States (75):
  - Univ. of Alabama Birmingham NICHD CRS (5096), Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Miller Children's Hospital Long Beach (5093), Long Beach, California
  - Los Angeles County Medical Center/USC, Los Angeles, California
  - Usc La Nichd Crs (5048), Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CR (3601), Los Angeles, California
  - Univ of California, San Diego (4601), San Diego, California
  - Univ. of California San Francisco NICHD CRS (5091), San Francisco, California
  - Harbor-UCLA Med Ctr (5045), Torrance, California
  - University of Colorado Denver NICHD CRS (5052), Denver, Colorado
  - Connecticut Childrens Medical Center (Pediatric), Farmington, Connecticut
  - University of Connecticut, Farmington, Farmington, Connecticut
  - Yale Univ School of Med, New Haven, Connecticut
  - Children's National Medical Center Washington DC NICHD CRS (5015), Washington D.C., District of Columbia
  - Washington Hospital Center NICHD CRS (5023), Washington D.C., District of Columbia
  - Howard Univ Hosp (5044), Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - South Florida CDC Ft Lauderdale NICHD CRS (5055), Fort Lauderdal, Florida
  - University of Florida Jacksonville (5051), Jacksonville, Florida
  - Jackson Memorial Hosp, Miami, Florida
  - University of Miami Pediatric/Perinatal HIV/AIDS (4201), Miami, Florida
  - University of South Florida at Tampa (5018), St. Petersburg, Florida
  - Med College of Georgia, Augusta, Georgia
  - The Medical Center, Columbus, Georgia
  - Womens & Childrens HIV Program, Chicago, Illinois
  - Mt Sinai Hosp Med Ctr / Dept of Pediatrics, Chicago, Illinois
  - Univ of Illinois, Chicago, Illinois
  - Cook County Hospital, Chicago, Illinois
  - Rush University Cook County Hospital NICHD CRS (5083), Chicago, Illinois
  - Chicago Childrens Memorial Hosp (Pediatric), Chicago, Illinois
  - Univ of Chicago Children's Hosp (4001), Chicago, Illinois
  - Tulane University New Orleans (5095), New Orleans, Louisiana
  - Tulane-Lakeside Hospital, New Orleans, Louisiana
  - Tulane University Charity Hosp of New Orleans (7201), New Orleans, Louisiana
  - University of Maryland Baltimore NICHD CRS (5094), Baltimore, Maryland
  - Johns Hopkins University NICHD CRS (5092), Baltimore, Maryland
  - Children's Hospital of Boston NICHD CRS (5009), Boston, Massachusetts
  - Boston Med Ctr (Pediatric) (5011), Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS (7301), Worcester, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Hutzel Hospital (5089), Detroit, Michigan
  - Wayne State University Detroit Children's Hosp of Michigan (5041), Detroit, Michigan
  - St. Louis Children's Hosp, St Louis, Missouri
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp (P2802), Newark, New Jersey
  - New Jersey Medical School (2802), Newark, New Jersey
  - Univ of Med & Dentistry of New Jersey/Univ Hosp, Newark, New Jersey
  - Children's Hospital at Downstate, Brooklyn, New York
  - New York University NY (5012), New York, New York
  - NYU/Bellevue Hospital, New York, New York
  - Metropolitan Hosp Ctr (5003), New York, New York
  - Columbia IMPAACT CRS (4101), New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - State Univ of New York at Stony Brook (5040), Stony Brook, New York
  - SUNY Upstate Medical Univ, Syracuse, New York
  - Lincoln Medical & Mental Health Center, The Bronx, New York
  - Bronx-Lebanon Hospital IMPAACT (6901), The Bronx, New York
  - Jacobi Med. Ctr. Bronx NICHD CRS (5013), The Bronx, New York
  - Montefiore Medical / AECOM, The Bronx, New York
  - Duke Univ (Pediatric) (DUMC) (4701), Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Hahnemann University Hospital (6706), Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Children's Hospital of Philadelphia (6701), Philadelphia, Pennsylvania
  - The Regional Med Ctr, Memphis (6502), Memphis, Tennessee
  - St. Jude Childrens Research Hosp, Memphis (6501), Memphis, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Texas Children's Hosp / Baylor Univ (3801), Houston, Texas
  - Univ of Washington Children's Hospital Seattle (5017), Seattle, Washington
  - Harborview Medical Center NICHD CRS (5027), Seattle, Washington
  - University of Washington NICHD CRS (5029), Seattle, Washington
- Puerto Rico (2):
  - University of Puerto Rico Pediatric HIV/AIDS (6601), San Juan
  - San Juan City Hosp. PR NICHD CRS (5031), San Juan

REFERENCES:
- [Background] Ciambrone D, Loewenthal HG, Bazerman LB, Zorilla C, Urbina B, Mitty JA. Adherence among women with HIV infection in Puerto Rico: the potential use of modified directly observed therapy (MDOT) among pregnant and postpartum women. Women Health. 2006;44(4):61-77. doi: 10.1300/j013v44n04_04. PMID 17456464
- [Background] Kingston MA, Letham CJ, McQuillan O. Adherence to antiretroviral therapy in pregnancy. Int J STD AIDS. 2007 Nov;18(11):787-9. doi: 10.1258/095646207782212216. PMID 18005515
- [Result] Bardeguez AD, Lindsey JC, Shannon M, Tuomala RE, Cohn SE, Smith E, Stek A, Buschur S, Cotter A, Bettica L, Read JS; PACTG 1025 Protocol Team. Adherence to antiretrovirals among US women during and after pregnancy. J Acquir Immune Defic Syndr. 2008 Aug 1;48(4):408-17. doi: 10.1097/QAI.0b013e31817bbe80. PMID 18614923
- [Derived] Momplaisir F, Hussein M, Kacanek D, Brady K, Agwu A, Scott G, Tuomala R, Bennett D. Perinatal Depressive Symptoms, Human Immunodeficiency Virus (HIV) Suppression, and the Underlying Role of Antiretroviral Therapy Adherence: A Longitudinal Mediation Analysis in the IMPAACT P1025 Cohort. Clin Infect Dis. 2021 Oct 20;73(8):1379-1387. doi: 10.1093/cid/ciab416. PMID 33982083
- [Derived] Jao J, Kacanek D, Williams PL, Geffner ME, Livingston EG, Sperling RS, Patel K, Bardeguez AD, Burchett SK, Chakhtoura N, Scott GB, Van Dyke RB, Abrams EJ; Pediatric HIV/AIDS Cohort Study and the International Maternal Pediatric Adolescent AIDS Clinical Trials P1025 Protocol; Pediatric HIV/AIDS Cohort Study and the International Maternal Pediatric Adolescent AIDS Clinical Trials P1025 Protocol. Birth Weight and Preterm Delivery Outcomes of Perinatally vs Nonperinatally Human Immunodeficiency Virus-Infected Pregnant Women in the United States: Results From the PHACS SMARTT Study and IMPAACT P1025 Protocol. Clin Infect Dis. 2017 Sep 15;65(6):982-989. doi: 10.1093/cid/cix488. PMID 28575201
- [Derived] Scott GB, Brogly SB, Muenz D, Stek AM, Read JS; International Maternal Pediatric Adolescent AIDS Clinical Trials Group (IMPAACT) P1025 Study Team. Missed Opportunities for Prevention of Mother-to-Child Transmission of Human Immunodeficiency Virus. Obstet Gynecol. 2017 Apr;129(4):621-628. doi: 10.1097/AOG.0000000000001929. PMID 28277349
- [Derived] Livingston EG, Huo Y, Patel K, Tuomala RE, Scott GB, Stek A; P1025 Team of the International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT) Group. Complications and Route of Delivery in a Large Cohort Study of HIV-1-Infected Women-IMPAACT P1025. J Acquir Immune Defic Syndr. 2016 Sep 1;73(1):74-82. doi: 10.1097/QAI.0000000000001021. PMID 27082506
- [Derived] Katz IT, Leister E, Kacanek D, Hughes MD, Bardeguez A, Livingston E, Stek A, Shapiro DE, Tuomala R. Factors associated with lack of viral suppression at delivery among highly active antiretroviral therapy-naive women with HIV: a cohort study. Ann Intern Med. 2015 Jan 20;162(2):90-9. doi: 10.7326/M13-2005. PMID 25599347